CLINICAL TRIAL: NCT01237431
Title: Importance of Liver Innervation for the Osmopressor Response in Humans
Acronym: HEP-Reflex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Jens Jordan, Medical School Hannover
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D-MHH-Hep_Reflex-EK5413
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2009-08

CONDITIONS: PHYSIOLOGICAL PHENOMENA
Keywords: Water drinking; osmoreceptors; autonomic failure; syncope; blood pressure; liver transplant
MeSH Terms: conditions — Pure Autonomic Failure; Syncope | interventions — Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- liver transplanted patients (Experimental): Target group to confirm the hypothesis. Transplantation has to be between 6 an 24 Month before participation.
  Interventions: Dietary Supplement: 500ml water intake
- kidney transplanted patients (Active Comparator): Control group, age, gender and medication matched. Transplantation has to be between 6 an 24 Month before participation.
  Interventions: Dietary Supplement: 500ml water intake

INTERVENTIONS:
Dietary Supplement: 500ml water intake — subjects have to ingest 500ml water within 5 minutes after resting 30 minutes in supine position

SUMMARY:
In patients with autonomic dysfunction water drinking elicits a pressor response mediated by sympathetic activation. If any, in healthy subjects there is only a slight increase in blood pressure. However, the sympathetic activation is observable by resting energy expenditure increases greater than 20%.

The investigators believe that the response to water may be mediated through sympathetic activation elicited by osmosensitve spinal afferents in the liver. Therefore, the investigators want to test water in liver transplant patients who have a denervated liver. Kidney transplant patients serve as control subjects. The investigators hypothesize that the increase in norepinephrine after water drinking is blunted in liver transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* 3 to 24 month past liver or kidney transplantation
* age 18 to 60
* written informed consent
* ability to understand the oral and written information

Exclusion Criteria:

* pregnancy or lactation
* transplantation of another organ
* chronic heart or vascular disease
* known alcohol or drug abuse
* psychiatric diseases (e.g. chronic depression, schizophrenia, drug addiction)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
norepinephrine plasma level | 30-40 minutes after water drinking

SECONDARY OUTCOMES:
pressure response | blood pressure 30-40 minutes after water drinking
  cardiovascular changes are monitored by finapress and ICG

CONTACTS AND LOCATIONS:
Locations (1):
- Hannover Medical School, Hanover, NDS, Germany

REFERENCES:
- [Derived] May M, Gueler F, Barg-Hock H, Heiringhoff KH, Engeli S, Heusser K, Diedrich A, Brandt A, Strassburg CP, Tank J, Sweep FC, Jordan J. Liver afferents contribute to water drinking-induced sympathetic activation in human subjects: a clinical trial. PLoS One. 2011;6(10):e25898. doi: 10.1371/journal.pone.0025898. Epub 2011 Oct 7. PMID 22016786